CLINICAL TRIAL: NCT05695508
Title: A Phase 2 Study to Evaluate Safety and Efficacy of Teclistamab-, Talquetamab-, and JNJ-79635322-based Combination Regimens in Participants With Newly Diagnosed Transplant Eligible Multiple Myeloma
Brief Title: GMMG-HD10 / DSMM-XX / 64007957MMY2003, MajesTEC-5
Acronym: HD10/DSMMXX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: Janssen Research & Development, LLC (Industry); Deutsche Studiengruppe Multiples Myelom (DSMM) (Unknown)
Responsible Party: Principal Investigator, Marc Raab, Prof. Dr. med., University of Heidelberg Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMMG-HD10/DSMM-XX
Record Dates: First submitted 2022-11-30; First posted 2023-01-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Focal Adhesion Protein-Tyrosine Kinases; daratumumab; Dexamethasone; Lenalidomide; Bortezomib; talquetamab

STUDY DESIGN:
Intervention Model Description: Induction phase contains 6 cycles of Tec-DRd [Arm A, A1, D] , Tec-DVRd [Arm B], Tal-DRd [Arm E, E1] or Tal-DVRd [Arm F, F1] or JNJ-79635322-DRd [Arm G] . Enrollment will be staggered with Arm A opening first.
  Induction therapy (except Arms D and G) is followed by HDT and a single ASCT according to local SoC. Participants will receive maintenance treatment with Tec-D [Arm A, A1, B, E. F] or Tal-D [E1, F1] or JNJ-79635322-D [Arm G].
  Arm C, C1 and C2 participants will enter the study at Maintenance Treatment with Tec-D or Tal-DR after induction, HDT, and ASCT according to local SoC (outside of the study).
  All Arms receive maintenance treatment for a max. of 18 cycles or until confirmed PD, death, intolerable toxicity, loss to follow-up, or consent withdrawal, whichever comes first. An optional EoT is possible for those patients who have sustained MRD negativity of 12 months.
  Periodic safety evaluations will be conducted to ensure that treatment is safe and tolerable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Arm A Tec-DRd Induction and Tec-D Maintenance (Experimental): Arm A participants will receive teclistamab as subcutaneous (SC) injection in combination with daratumumab SC, lenalidomide and dexamethasone in 6 cycles of induction therapy, followed by teclistamab SC injection in combination with daratumumab SC in maximum 18 cycles of maintenance therapy.
  Interventions: Drug: Teclistamab (Tec); Drug: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide
- Arm B Tec-DVRd Induction and Tec-D Maintenance (Experimental): Arm B participants will receive teclistamab as subcutaneous (SC) injection in combination with daratumumab SC, lenalidomide, dexamethasone and bortezomib in 6 cycles of induction therapy, followed by teclistamab SC injection in combination with daratumumab SC in maximum 18 cycles of maintenance therapy.
  Interventions: Drug: Teclistamab (Tec); Drug: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Bortezomib
- Arm C Tec-D Maintenance (Experimental): Arm C participants will receive maximum 18 cycles of teclistamab SC injection in combination with daratumumab SC and lenalidomide as maintenance therapy.
  Interventions: Drug: Teclistamab (Tec); Drug: Daratumumab
- Arm A1 Tec-DRd Induction and Tec-D Maintenance (Experimental): Arm A1 participants will receive teclistamab as subcutaneous (SC) injection in combination with daratumumab SC, lenalidomide and dexamethasone in 6 cycles of induction therapy, followed by teclistamab SC injection in combination with daratumumab SC in maximum 18 cycles of maintenance therapy.
  Interventions: Drug: Teclistamab (Tec); Drug: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide
- Arm C2 Tal-DR Maintenance (Experimental): Arm C2 participants will receive maximum 18 cycles of talquetamab SC injection in combination with daratumumab SC and lenalidomide as maintenance therapy.
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Talquetamab
- Arm D Tec-DRd Induction and Tec-Tal following induction (Experimental): Arm D participants will receive teclistamab as subcutaneous (SC) injection in combination with daratumumab SC, lenalidomide and dexamethasone in 6 cycles of induction therapy, followed by a combination of teclistamab and talquetamab SC injection in maximum 18 cycles of following induction therapy.
  Interventions: Drug: Teclistamab (Tec); Drug: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Talquetamab
- Arm E Tal-DRd Induction and Tec-D Maintenance (Experimental): Arm E participants will receive talquetamab as subcutaneous (SC) injection in combination with daratumumab SC, lenalidomide and dexamethasone in 6 cycles of induction therapy, followed by teclistamab SC injection in combination with daratumumab SC in maximum 18 cycles of maintenance therapy.
  Interventions: Drug: Teclistamab (Tec); Drug: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Talquetamab
- Arm E1 Tal-DRd Induction and Tal-D Maintenance (Experimental): Arm E1 participants will receive talquetamab as subcutaneous (SC) injection in combination with daratumumab SC, lenalidomide and dexamethasone in 6 cycles of induction therapy, followed by talquetamab SC injection in combination with daratumumab SC in maximum 18 cycles of maintenance therapy.
  Interventions: Drug: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Talquetamab
- Arm F Tal-DVRd Induction and Tec-D Maintenance (Experimental): Arm F participants will receive talquetamab as subcutaneous (SC) injection in combination with daratumumab SC, bortezomib, lenalidomide and dexamethasone in 6 cycles of induction therapy, followed by teclistamab SC injection in combination with daratumumab SC in maximum 18 cycles of maintenance therapy.
  Interventions: Drug: Teclistamab (Tec); Drug: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Bortezomib; Drug: Talquetamab
- Arm F1 Tal-DVRd Induction and Tal-D Maintenance (Experimental): Arm F1 participants will receive talquetamab as subcutaneous (SC) injection in combination with daratumumab SC, bortezomib, lenalidomide and dexamethasone in 6 cycles of induction therapy, followed by talquetamab SC injection in combination with daratumumab SC in maximum 18 cycles of maintenance therapy.
  Interventions: Drug: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Bortezomib; Drug: Talquetamab
- Arm-G JNJ-79635322-DRd induction - JNJ-79635322-D following ind (Experimental): Arm G participants will receive six 28-day cycles of JNJ-79635322-DRd induction, followed byJNJ-79635322-D treatment for a maximum of eighteen 28-day cycles or until confirmed PD, death, intolerable toxicity, loss to follow-up, or consent withdrawal, whichever comes first. Tec-Tal or JNJ-79635322-D treatment can be discontinued when 12 months of sustained MRD negativity has been observed during the study.
  Interventions: Drug: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: JNJ-79635322

INTERVENTIONS:
Drug: Teclistamab (Tec) — Subcutaneous administration of Teclistamab
  Other Names: JNJ-64007957
  Arms: Arm A Tec-DRd Induction and Tec-D Maintenance; Arm A1 Tec-DRd Induction and Tec-D Maintenance; Arm B Tec-DVRd Induction and Tec-D Maintenance; Arm C Tec-D Maintenance; Arm D Tec-DRd Induction and Tec-Tal following induction; Arm E Tal-DRd Induction and Tec-D Maintenance; Arm F Tal-DVRd Induction and Tec-D Maintenance
Drug: Daratumumab — Subcutaneous administration of Daratumumab
Drug: Dexamethasone — administered i.v. or orally
  Arms: Arm A Tec-DRd Induction and Tec-D Maintenance; Arm A1 Tec-DRd Induction and Tec-D Maintenance; Arm B Tec-DVRd Induction and Tec-D Maintenance; Arm D Tec-DRd Induction and Tec-Tal following induction; Arm E Tal-DRd Induction and Tec-D Maintenance; Arm E1 Tal-DRd Induction and Tal-D Maintenance; Arm F Tal-DVRd Induction and Tec-D Maintenance; Arm F1 Tal-DVRd Induction and Tal-D Maintenance; Arm-G JNJ-79635322-DRd induction - JNJ-79635322-D following ind
Drug: Lenalidomide — Administration oral
  Arms: Arm A Tec-DRd Induction and Tec-D Maintenance; Arm A1 Tec-DRd Induction and Tec-D Maintenance; Arm B Tec-DVRd Induction and Tec-D Maintenance; Arm C2 Tal-DR Maintenance; Arm D Tec-DRd Induction and Tec-Tal following induction; Arm E Tal-DRd Induction and Tec-D Maintenance; Arm E1 Tal-DRd Induction and Tal-D Maintenance; Arm F Tal-DVRd Induction and Tec-D Maintenance; Arm F1 Tal-DVRd Induction and Tal-D Maintenance; Arm-G JNJ-79635322-DRd induction - JNJ-79635322-D following ind
Drug: Bortezomib — Subcutaneous administration
  Arms: Arm B Tec-DVRd Induction and Tec-D Maintenance; Arm F Tal-DVRd Induction and Tec-D Maintenance; Arm F1 Tal-DVRd Induction and Tal-D Maintenance
Drug: Talquetamab — Subcutaneous administration of Daratumumab
  Arms: Arm C2 Tal-DR Maintenance; Arm D Tec-DRd Induction and Tec-Tal following induction; Arm E Tal-DRd Induction and Tec-D Maintenance; Arm E1 Tal-DRd Induction and Tal-D Maintenance; Arm F Tal-DVRd Induction and Tec-D Maintenance; Arm F1 Tal-DVRd Induction and Tal-D Maintenance
Drug: JNJ-79635322 — Subcutaneous administration
  Arms: Arm-G JNJ-79635322-DRd induction - JNJ-79635322-D following ind

SUMMARY:
A Phase 2 Study to Evaluate Safety and Efficacy of Teclistamab-, Talquetamab-, and JNJ-79635322-based Combination Regimens in Participants with Newly Diagnosed Transplant Eligible Multiple Myeloma

OBJECTIVES:

To evaluate the safety and tolerability of teclistamab-, talquetamab-, and JNJ-79635322-based combination regimens over the entire treatment phase for each arm, in participants with ND-TEMM

To evaluate the efficacy of teclistamab- and talquetamab-based combination regimens as induction and post-transplant maintenance treatments; JNJ-79635322-based combinations as induction and as replacement for HDT+ASCT following induction; and teclistamab in combination with talquetamab

DETAILED DESCRIPTION:
OVERALL DESIGN:

160 participants will be enrolled with 10 participants in Arm A, 20 participants in Arm A1, 20 participants in Arm B, 10 participants in Arms C and 10 in C2, 20 participants in Arm D, 10 participants in each Arm E, E1 and optionally F and F, and 20 participants in Arm G. Cohorts may be further expanded.

Arms A, A1, B, D, E, E1, F, F1 will receive Induction therapy of 6 cycles (28-days each):

Treatment: Tec-DRd (Arm A, A1), Tec-DVRd (Arm B), Tal-DRd (Arms E, E1), Tal-DVRd (Arms F, F1) followed by HDT and a single ASCT according to local SoC treatment. Thereafter a Maintenance Therapy of maximum 18 cycles with either Tec-D (Arms A, A1, B, E, F) or Tal-D (E1, F1) is performed.

Arm D will receive 6 28-days cycles Tec-DVRd induction followed by 18 cycles Tec-Tal. Arm G will receive 6 28-day cycles of JNJ-79635322-DRd induction, followed by JNJ-79635322-D. No HDT ASCT will be performed in Arm D and Arm G.

In Arm C and C2 participants will enter the study for maintenance treatment of 18 cycles with Tec-D (Arm C) or Tal-DR (Arm C2) , after induction, HDT and ASCT according to local SoC (outside of the study).

Participants will receive maintenance treatment or following induction treatment (Arm D and G) for a maximum of 18 cycles or until confirmed progressive disease, death, intolerable toxicity, loss to follow-up, or consent withdrawal, whichever comes first. An optional end of treatment is possible for patients who have 12 months sustained MRD negativity.

Periodic safety evaluations will be conducted to ensure that treatment is safe and tolerable. Upon treatment discontinuation, an EOT Visit will be conducted. Thereafter, the participant will continue in the Follow-up Phase until death, withdrawal of consent, loss to follow-up, or end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

- 18 years of age to 70 years of age, inclusive

* Have an ECOG performance status score of 0 to 2 at screening
* Have an ECOG performance status score of 0 to 2 at screening and immediately prior to the start of administration of study treatment

Participants in Arms A, A1, B, D, E, E1, F, F1 and G must also satisfy all of the following criteria to be enrolled in the study:

1. Documented multiple myeloma requiring treatment as defined by the criteria below:

1. Multiple myeloma diagnosis according to the IMWG diagnostic criteria
2. Measurable disease at screening as defined by any of the following:

   1. Serum M-protein level ≥1.0 g/dL or 2. Urine M-protein level ≥200 mg/24 hours or 3. Serum immunoglobulin free light chain level ≥10 mg/dL and abnormal serum free light chain ratio 2. Newly diagnosed participants for whom HDT and ASCT is part of the intended treatment plan (except Arm D and G participants).

   Participants Arm C and C2 must also satisfy all of the following criteria:
   1. Newly diagnosed multiple myeloma according to IMWG criteria.
   2. Must have received 4 to 6 28-day cycles of 3 or 4 drug-induction therapy that includes a proteasome inhibitor and/or an IMiD with or without anti-CD38 monoclonal antibody and a single or tandem ASCT. Post-ASCT consolidation is permitted for up to 2 cycles as long as the total number of induction plus consolidation cycles does not exceed 6.

   3 Must have received only one line of therapy and achieved at least a PR as per IMWG 2016 response criteria based on the investigator's assessment. Participants with plasmacytomas at the time of diagnosis must meet IMWG 2016 response criteria for ≥PR based on repeat imaging utilizing the same modality 4. Must have received HDT and ASCT within 12 months of the start of induction therapy and be within 6 months of the last ASCT (7 months for participants who received consolidation) at the time of enrollment.

   Exclusion Criteria:

   - CNS involvement or clinical signs of meningeal involvement of multiple myeloma.

   - Stroke or seizure within 6 months prior study start Cycle1 Day1.

   - History of transplantations requiring immunosuppressive therapy.

   - Seropositive for HIV, HEP B, Active Hep C infection (details see protocol).

   - COPD with a FEV1 <50% of predicted normal.

   - Moderate /severe persistent asthma within the past 2 years or any uncontrolled asthma. Exclude if FEV1 <50% of predicted normal.

   - Concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures, or that in the investigators opinion would constitute a hazard for participants.

   - Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug/excipients.

   - Pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of any study treatment regimen.

   - Plans to father a child while enrolled in this study or within 100 days after the last dose of any component of the study treatment regimen.

   Arm A, A1, B, D, E, E1, F, F1
   * Prior or current systemic therapy or stem cell transplant for any plasma cell dyscrasia, with the exception of emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment.
   * Arm B only: Peripheral neuropathy or neuropathic pain Grade 2 or higher as defined by the NCI-CTCAE Version 5.

   Due to a potential interaction with bortezomib, received a strong CYP3A4 inducer within 5 half-lives prior to enrollment

   Arm C and C2

   - Discontinued treatment due to any AE related to lenalidomide as determined by the investigator.
   * Progressed on multiple myeloma therapy at any time prior to screening.
   * Received a cumulative dose of corticosteroids equivalent to ≥40 mg of dexamethasone within the 14 day period before the start of study treatment administration.
   * Intolerant to the starting dose of lenalidomide (10 mg).

   For further details on inclusion/exclusion criteria please refer to the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
number of incidence and severity of adverse events [safety and tolerability] | through study completion, up to 28 months

SECONDARY OUTCOMES:
MRD negativity rate | after 6 cycles (each cycle is 28 days) induction therapy (app.month 6), after High Dose Therapy (app. month 10), after 18 cycles (each cycle is 28 days) of maintenance therapy (app. month 28)
  MRD negativity rate measured by Flow Cytometry
Response on therapy [efficacy] | after each cycle (each cycle is 28 days) induction ( app. at month 1,2,...,6), after High Dose therapy (app. month 10), after each cycle (each cycle is 28 days) of maintenance (app. at month 11,12, ...28), during FU every 3 months (app. up to 3-4 years)
  Response on therapy according to IMWG:
  * Overall Response Rate (ORR) (at least a PR or better)
  * Complete Response (CR) or better
  * Very Good Partial Response (VGPR) or better
  * Duration of Response (DoR)
Progression Free Survival [efficacy] | From randomization to the date of disease progression to death (app. up to 3-4 years)
Serum concentration of teclistamab, talquetamab and daratumumab [pharmacokinetics] | through study completion, up to 28 months
Presence of ADAs to teclistamab, talquetamab and daratumumab [immunogenicity] | through study completion, up to 28 months
Stem cell yield | after High Dose Therapy (after app. 10 months)
  feasibility of successful transplantation
days to engraftment | after High Dose Therapy (after app. 10 months)
  feasibility of successful transplantation

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (11):
  - Charité University Medicin Berlin, Berlin
  - Clinic Chemnitz gGmbH, Chemnitz
  - University Clinic Technical University Dresden, Dresden
  - University Clinic Düsseldorf, Düsseldorf
  - University Clinic Freiburg, Freiburg im Breisgau
  - Hamburg University Clinic Eppendorf, Hamburg
  - Asklepios Clinic Hamburg Altona, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - University Clinic Schleswig-Holstein Campus Kiel, Kiel
  - Technical University Munich, Munich
  - University Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No